CLINICAL TRIAL: NCT01597973
Title: Randomized Controlled Trial for the Treatment of Extensively Drug-Resistant Gram-negative Bacilli (OVERCOME)
Brief Title: Trial for the Treatment of Extensively Drug-Resistant Gram-negative Bacilli (OVERCOME)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, keith kaye, Keith Kaye, M.D.,M.P.H Study PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIH 10-0065
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pneumonia; Blood Stream Infection
MeSH Terms: conditions — Pneumonia | interventions — Colistin; Meropenem; colistinmethanesulfonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colistin and meropenem (Active Comparator)
  Interventions: Drug: colistin and meropenem
- colistin and placebo (Active Comparator)
  Interventions: Drug: colistin and placebo

INTERVENTIONS:
Drug: colistin and meropenem — colistin standard loading dose, maintenance dose based on patients renal function meropenem- dose based on patients renal function
  Other Names: Colistimethate; Meropenem
  Arms: colistin and meropenem
Drug: colistin and placebo — colistin- loading dose standard, maintenance dosed based on patients renal function placebo- mimic meropenem (blinded)
  Other Names: Colistimethate
  Arms: colistin and placebo

SUMMARY:
Approximately 444 subjects who are greater than or equal to 18 to 95 years of age, are non-pregnant, and are in the inpatient setting of one of the study sites will be evaluated to treatment efficacy. Analysis will include subjects with bloodstream infection (BSI) or pneumonia due to at least one of the following gram-negative bacilli organisms: Acinetobacter baumannii, Klebsiella spp, Escherichia coli, Enterobacter spp. and/or Pseudomonas aeruginosa that demonstrates in vitro non-susceptibility defined as extensively drug-resistant Gram-negative bacilli (XDR-GNB) which includes XDR-AB, XDR-PA and CRE. If a subject has both BSI and pneumonia at the time of study enrollment, they will be included as a subject with pneumonia.

Objectives:

Primary:

•Determine whether the treatment regimen of Colistimethate sodium (colistin) combined with a carbapenem (imipenem or meropenem) is associated with a decreased risk for mortality compared to colistin alone for subjects with bloodstream infection (BSI) and/or pneumonia due to XDR-GNB.

Secondary:

•Determine what treatment regimen (colistin monotherapy or colistin combined with a carbapenem (imipenem or meropenem) is more likely to reduce the emergence of colistin resistance among XDR-GNB isolates during therapy.

DETAILED DESCRIPTION:
The Gram-negative bacilli organisms Acinetobacter baumannii, Klebsiella spp., Escherichia coli, Enterobacter spp. and Pseudomonas aeruginosa have become a frequent cause of bloodstream infection and pneumonia in the hospital and other healthcare settings. Among these pathogens, antimicrobial resistance has emerged to many classes of antimicrobial agents. Most concerning, has been the emergence of resistance to group 2 carbapenems (such as imipenem). In several regions of the world, including Southeastern Michigan, strains of extensively-drug resistant Gram-negative bacilli (XDR-GNB) that exhibit resistance to most, and in some cases all types of available antimicrobial agents, including group 2 carbapenems, have emerged and disseminated. Treatment options for XDR-GNB typically include Colistimethate sodium (referred to as colistin in this study), used alone (monotherapy) or in combination with other agents. Unfortunately, resistance to colistin has begun to emerge in some strains of XDR-GNB, which is a truly concerning development, since colistin is one of the last remaining treatment options for XDR-GNB. No prospective, randomized controlled trials have been conducted to evaluate the clinical efficacy of colistin monotherapy versus colistin-containing combination therapy or the impact of these therapeutic modalities on the emergence of colistin resistance among XDR-GNB. We plan to conduct a double-blind randomized controlled trial including patients with pneumonia and bloodstream infection due to XDR-GNB. After enrollment, subjects will be randomized to receive 14 days of either colistin monotherapy or colistin plus meropenem.

In the Detroit metro area, infections due to XDR-GNB have developed into a regional challenge and common problem. We have assembled a multi-disciplinary team that includes Infectious Diseases researchers, clinicians, infectious diseases pharmacists, microbiologists, epidemiologists and statistical experts to address critically important questions and challenges regarding the management of bloodstream infection and pneumonia due to XDR-GNB. Specifically, we hypothesize that the combination of colistin and imipenem will provide superior efficacy in the treatment of XDR-GNB pneumonia and bloodstream infection and will prevent the emergence of decreased susceptibility to colistin among XDR-GNB strains. We also aim to analyze tools that could be used in "real time" to aid clinicians treating patients with infection due to XDR-GNB. For example, we aim to analyze the association between the presence of in vitro synergy of the colistin and carbapenem (imipenem or meropenem) combination (as determined by E-test) and clinical outcomes; and the association between colistin plasma levels and clinical outcomes and the development of nephrotoxicity.

Due to the growing threat of XDR-GNB around the world, several international sites were subsequently added including sites in Asia, Israel, and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Adults (> 18 years to 95 years of age), at one of the study sites.
* Diagnosis of BSI and/or pneumonia due to a preliminary result of gram-negative non-lactose fermenter that is oxidase negative; or a final results of XDR-A. baumannii; carbapenem-resistant Enterobacteriaceae; or XDR- P. aeruginosa and/or patients with suspected BSI and/or HAP (hospital acquired pneumonia) and who have had a prior history (within last 6 months) of XDR-GNB that was susceptible to colistin.

  o If final results do not indicate that the pathogen is an XDR-GNB, and identifies alternative treatment options, the patient would be eligible for the study if the subject is allergic to all the alternative treatment options.
* Patients with polymicrobial respiratory or blood infections, including XDR-GNB and one or more pathogens, will be included in the study, as long as the XDR-GNB is determined to be a true pathogen (AB, CRE or PA). Other pathogens will be treated with antimicrobial agents as determined by the treating physician.
* If more than one XDR-GNB study pathogens is identified as a study pathogen causing BSI and/or pneumonia, then the first study pathogen recovered will be considered as the primary study pathogen. If more than one study pathogen is recovered from the same culture, then the infection will be categorized as being caused by multiple study pathogens.
* Patients with a life expectancy of > 24 hours
* Signed written informed consent and HIPAA Authorization form (US sites)

Exclusion Criteria:

* Female patients who are pregnant
* Female patients who are nursing
* Patients who are prisoners
* Patients who are less than 18 years of age or greater than or equal to 96 years of age
* Patients with neutropenia (WBC < 500 cells/mm3)
* The presence of any of the following known clinical syndromes involving XDR-GNB as a pathogen which necessitate durations of antimicrobial therapies greater than 14 days: endocarditis, osteomyelitis, prosthetic joint infections, meningitis and/or other central nervous system infections.
* Patients receiving valproic acid (with or without a known seizure disorder).
* Patients who received 72 hours or more of polymyxin treatment (intravenous or inhaled [pneumonia]) within 96 hours of enrollment.
* Patients who have end-stage renal disease requiring hemodialysis, will be excluded from evaluation pertaining to nephrotoxicity in the per protocol population.
* Patients with known Type 1 or other severe drug allergy to either of the study drugs or to β-lactams.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2012-10-06 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2020-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith S Kaye, MD, MPH, Principal Investigator — University of Michigan
Locations (19):
- United States (6):
  - Jackson Memorial Hospital-Jackson Health System, Miami, Florida
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - Mount Sinai Hospital, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Bulgaria
- Greece (5):
  - University Hospital of Heraklion, Crete, Crete
  - Evangelismos General Hospital of Athens, Athens
  - General Hospital of Athens "Laiko" 1st Department of Medicine, Athens
  - Attikon University General Hospital of Athens, Athens
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Israel (4):
  - Assaf Harofeh Medical Center, Ẕerifin, Beer Yaakov
  - Rabin Medical Centre, Beilinson Campus, Petah Tikva, Central District
  - Rambam Health Care Campus, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Universita della Campania 'Luigi Vanvitelli', Naples, Italy
- Chang Gung Memorial Hospital, Taoyuan District, Kwei-San, Taiwan
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Derived] Kaye KS, Marchaim D, Thamlikitkul V, Carmeli Y, Chiu CH, Daikos G, Dhar S, Durante-Mangoni E, Gikas A, Kotanidou A, Paul M, Roilides E, Rybak M, Samarkos M, Sims M, Tancheva D, Tsiodras S, Kett D, Patel G, Calfee D, Leibovici L, Power L, Munoz-Price S, Stevenson K, Susick L, Latack K, Daniel J, Chiou C, Divine GW, Ghazyaran V, Pogue JM. Colistin Monotherapy versus Combination Therapy for Carbapenem-Resistant Organisms. NEJM Evid. 2023 Jan;2(1):10.1056/evidoa2200131. doi: 10.1056/evidoa2200131. Epub 2022 Dec 6. PMID 37538951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 467 participants completed an informed consent document, 3 were deemed ineligible
Groups:
- Colistin and Placebo: colistin and placebo: colistin- loading dose standard, maintenance dosed based on patient's renal function placebo- mimic meropenem (blinded)
- Colistin and a Carbapenem: colistin and a carbapenem: colistin standard loading dose, maintenance dose based on patient's renal function carbapenem- dose based on patient's renal function
Period: Overall Study
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Started (Started means randomized, here.) | 234 | 230
Began First Dose | 230 | 228
Completed | 214 | 211
Not Completed | 20 | 19
Not completed — Found ineligible before study medication started | 4 | 2
Not completed — Eligible pathogen not confirmed | 14 | 15
Not completed — LAR not authorized to consent | 0 | 1
Not completed — Ineligible due to early seizures | 1 | 0
Not completed — Ineligible due to non-target infection | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem | Total
Number analyzed (Participants) | 234 | 230 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (16.3) | 68.4 (15.4) | 68.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 84 | 174
  Male | 144 | 146 | 290
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 96 | 91 | 187
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 14 | 31
  White | 116 | 120 | 236
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Greece | 14 | 15 | 29
  United States | 26 | 23 | 49
  Taiwan | 29 | 28 | 57
  Italy | 4 | 5 | 9
  Israel | 89 | 93 | 182
  Thailand | 68 | 64 | 132
  Bulgaria | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Determine whether the treatment regimen of colistin combined with a carbapenem (imipenem or meropenem) is associated with a decreased risk for all-cause mortality during the 30 day post-enrollment period compared to colistin combined with a placebo for subjects with bloodstream infection (BSI) and/or pneumonia due to extensively drug-resistant Gram-negative bacilli (XDR-GNB).
Time Frame: participants will be followed daily for the duration of hospital stay, an expected average of 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Colistin and Placebo: colistin and placebo: colistin- loading dose standard, maintenance dose based on patient's renal function placebo- mimic meropenem (blinded)
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Number analyzed (Participants) | 214 | 211
Participants
  Dead | 92 | 78
  Alive | 122 | 133
Statistical Analysis 1: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Test type: Superiority; p = 0.21, Chi-squared

2. Secondary Outcome: Number of Participants Who Develop Colistin Resistance
Description: Determine what treatment regimen (colistin monotherapy (combined with placebo)) or colistin combined a carbapenem (imipenem or meropenem) is more likely to reduce the frequency of emergence of colistin resistance among XDR-GNB isolates during therapy. Measurements of Minimum Inhibitory Concentration of colistin to XDR-GNB. This is shown below as numbers of those subjects who develop colistin resistance and their percentages of the total completed population.
Time Frame: patients' resistance data will be collected up to 30 days
Population: Follow up cultures were unable to be obtained for some subjects. Therefore emergence of resistance status for those subjects could not be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Number analyzed (Participants) | 173 | 173
Participants | 18 | 15
Statistical Analysis 1: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Test type: Superiority; p = 0.5830, Chi-squared

3. Secondary Outcome: Clinical Failure at the End of Therapy
Description: Clinical failure as defined by either Blood Stream Infection (BSI) or Pneumonia; based on death between 48 hours and end of treatment, medication change from protocol, a positive blood culture after 5 days of blood stream infection treatment, or no improvements in PaO2/FiO2 at end of treatment.
Time Frame: 48 hours after end of treatment, that is up to 16 days
Population: 54 patients were omitted due to death before 48 hours (n=40) or incomplete PaO2/FiO2 data (n=14).
Measure: Count of Participants; unit: Participants
Groups:
- Colistin and Placebo: colistin and placebo: colistin- loading dose standard, maintenance dosed based on patient's renal function placebo-mimic meropenem (blinded)
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Number analyzed (Participants) | 186 | 185
Participants | 115 | 97
Statistical Analysis 1: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Test type: Superiority; p = 0.07, Chi-squared

4. Secondary Outcome: Microbiologic Cure at the End of Therapy
Description: Microbiologic cure at the end of therapy as defined by the number of participants who no longer have the causative XDR-GNB pathogens for their BSI or pneumonia identified based on microbiologic testing
Time Frame: From 5 days after enrollment up to 14 days following enrollment (i.e. end of treatment)
Population: Some patients did not have data in the time window of interest (from 5 days following enrollment until end of treatment, 14 days) (e.g. from some specimens not being produced or available).
Measure: Count of Participants; unit: Participants
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Number analyzed (Participants) | 169 | 174
Participants
  Cure | 112 | 105
  Failure | 57 | 69
Statistical Analysis 1: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Test type: Superiority; p = 0.255, Chi-squared

5. Secondary Outcome: Number of Participants With Toxicities Related to Treatment Medications
Description: Frequency is shown for each of the following: Nephrotoxicity, Hepatotoxicity, Seizures, Neurotoxicity, Hypersensitivity reaction
Time Frame: Up to 16 days
Population: Follow up creatinine clearance data was missing from many patients resulting in a smaller analysis population for nephrotoxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
Number analyzed (Participants) | 214 | 211
Participants
  Nephrotoxicity: number analyzed (Participants) | 170 | 174
  Nephrotoxicity | 88 | 85
  Hypersensitivity reaction | 3 | 7
  Hepatotoxicity | 32 | 31
  Seizures | 4 | 3
  Neurotoxicity | 11 | 5
Statistical Analysis 1: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; nephrotoxicity analysis; Test type: Superiority; p = 0.59, Chi-squared
Statistical Analysis 2: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Hypersensitivity analysis; Test type: Superiority; p = 0.22, Fisher Exact
Statistical Analysis 3: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Hepatoxicity analysis; Test type: Superiority; p = 0.94, Chi-squared
Statistical Analysis 4: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Seizures analysis; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 5: Comparison: Colistin and Placebo vs Colistin and a Carbapenem; Neurotoxicity analysis; Test type: Superiority; p = 0.20, Fisher Exact

ADVERSE EVENTS:
Time Frame: For AEs, the assessment period begins at the time of enrollment and continues until 48 hours after end of treatment, that is up to 16 days. (as 48 hours is total removal of colistin from the patient has occurred). All-Cause Mortality, the Primary Objective is assessed up to 30 days after enrollment.
Groups:
- Colistin and a Carbapenem: colistin and carbapenem: colistin standard loading dose, maintenance dose based on patient's renal function carbapenem- dose based on patient's renal function
Arm/Group | Colistin and Placebo | Colistin and a Carbapenem
All-Cause Mortality (participants affected / at risk) | 98/230 | 85/228
Serious Adverse Events (participants affected / at risk) | 13/230 | 10/228
Other Adverse Events (participants affected / at risk) | 169/230 | 161/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colistin and Placebo (N=230) | Colistin and a Carbapenem (N=228)
Abdominal infection (Infections and infestations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Intestinal ischemia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Progression of pre-existing cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Seizure (Nervous system disorders) | 3 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colistin and Placebo (N=230) | Colistin and a Carbapenem (N=228)
ALT increased (Investigations) | 3 | 7
APTT increased (Investigations) | 0 | 1
AST increased (Investigations) | 2 | 2
AV block first degree (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain generalised (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Abnormal ECG (Investigations) | 2 | 0
Abnormal EEG (Investigations) | 1 | 0
Abnormal arterial blood gases (Investigations) | 6 | 2
Above knee amputation (Surgical and medical procedures) | 0 | 1
Absolute lymphocyte count decreased (Investigations) | 1 | 1
Absolute lymphocyte count increased (Investigations) | 1 | 2
Absolute monocyte count increased (Investigations) | 2 | 1
Absolute neutrophil count increased (Investigations) | 2 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Acinetobacter baumannii test positive (Investigations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Activated partial thromboplastin time increased (Investigations) | 3 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Acute bronchitis (Infections and infestations) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 78 | 69
Acute pain (General disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0
Alanine aminotransferase (Investigations) | 0 | 1
Alanine aminotransferase decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 2
Albumin globulin ratio decreased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 8 | 3
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Anasarca (General disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 12 | 6
Anion gap decreased (Investigations) | 1 | 0
Anisocoria (Eye disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Arterial blood pH increased (Investigations) | 1 | 0
Aspartate aminotransferase increase (Investigations) | 13 | 10
Aspartate aminotransferase increased (Investigations) | 8 | 9
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asystole (Cardiac disorders) | 1 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 | 0
BUN decreased (Investigations) | 2 | 1
Bacteria urine identified (Investigations) | 2 | 2
Band neutrophil count increased (Investigations) | 3 | 3
Bed sore (Skin and subcutaneous tissue disorders) | 1 | 0
Bedridden (Social circumstances) | 0 | 1
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bilirubin increased (Investigations) | 0 | 1
Bilirubin total decreased (Investigations) | 0 | 1
Bilirubin total increased (Investigations) | 1 | 3
Blistering (Skin and subcutaneous tissue disorders) | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood amylase decreased (Investigations) | 1 | 0
Blood bicarbonate increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 13 | 9
Blood carbon dioxide decreased (Investigations) | 2 | 0
Blood carbon dioxide increased (Investigations) | 0 | 3
Blood chloride decreased (Investigations) | 1 | 2
Blood chloride increased (Investigations) | 2 | 3
Blood eosinophils (Investigations) | 1 | 0
Blood eosinophils increased (Investigations) | 2 | 2
Blood gases abnormal (Investigations) | 1 | 1
Blood in urine (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 8 | 3
Blood lactic acid increased (Investigations) | 1 | 0
Blood myoglobin increased (Investigations) | 1 | 0
Blood pH decreased (Investigations) | 3 | 1
Blood pH increased (Investigations) | 2 | 0
Blood phosphorus increased (Investigations) | 2 | 1
Blood pressure diastolic decreased (Investigations) | 8 | 2
Blood pressure diastolic increased (Investigations) | 1 | 0
Blood pressure systolic decreased (Investigations) | 1 | 0
Blood prolactin abnormal (Investigations) | 1 | 0
Blood transfusion (Surgical and medical procedures) | 0 | 1
Blood urea nitrogen increased (Investigations) | 4 | 3
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1 | 0
Body temperature decrease (Investigations) | 2 | 2
Body temperature decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 2
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial mucus plug (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
C.difficile diarrhea (Infections and infestations) | 1 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Calcium ionized decreased (Investigations) | 1 | 1
Carbon dioxide decreased (Investigations) | 2 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Cardiac troponin T increased (Investigations) | 0 | 1
Cellulitis of arm (Infections and infestations) | 1 | 0
Central line placement (Surgical and medical procedures) | 1 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 1
Chemotherapy (Surgical and medical procedures) | 0 | 1
Chest tube insertion (Surgical and medical procedures) | 0 | 1
Chloride serum increased (Investigations) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholesterol blood decreased (Investigations) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Clostridium difficile test positive (Investigations) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Copper decreased (Investigations) | 0 | 1
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatine increased (Investigations) | 0 | 1
Creatinine decreased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 54 | 46
Creatinine urine decreased (Investigations) | 1 | 0
Crystal urine present (Investigations) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Delirium tremens (Psychiatric disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Dialysis device insertion (Surgical and medical procedures) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 2
Digoxin level increased (Investigations) | 1 | 0
Direct bilirubin increased (Investigations) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0
Drug fever (General disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Edema limbs (General disorders) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Elevated liver enzyme levels (Investigations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
End stage renal disease (ESRD) (Renal and urinary disorders) | 2 | 1
Endotracheal intubation (Surgical and medical procedures) | 0 | 1
Enlarged prostate (Reproductive system and breast disorders) | 0 | 1
Enlargement heart (Cardiac disorders) | 0 | 1
Enterococcus test positive (Investigations) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Eosinophil percentage increased (Investigations) | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Esophageal perforation (Gastrointestinal disorders) | 0 | 1
Febrile reaction (General disorders) | 1 | 0
Fecal occult blood (Investigations) | 0 | 1
Ferritin increased (Investigations) | 2 | 0
Fever (General disorders) | 4 | 4
Foley catheter (Surgical and medical procedures) | 0 | 1
GFR decreased (Investigations) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ischemia (Gastrointestinal disorders) | 0 | 1
General body pain (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 0 | 1
Generalized itching (Skin and subcutaneous tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Glucose urine abnormal (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
HDL cholesterol decreased (Investigations) | 1 | 0
HDL cholesterol increased (Investigations) | 1 | 0
HDL decreased (Investigations) | 1 | 0
Haptoglobin high (Investigations) | 1 | 1
HbA1C increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hematocrit decreased (Investigations) | 0 | 1
Hematuria (Renal and urinary disorders) | 3 | 4
Hemiplegia (Nervous system disorders) | 0 | 1
Hemodialysis (Surgical and medical procedures) | 0 | 1
Hemodynamic instability (Vascular disorders) | 0 | 1
Hemoglobin decreased (Investigations) | 0 | 2
Hepatitis A antibody positive (Investigations) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperchloremia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 4 | 4
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 | 2
Hypertension (Vascular disorders) | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglobulinemia (Blood and lymphatic system disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 11 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 5
Hyponatremia (Metabolism and nutrition disorders) | 7 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 3
Hypothermia (General disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
INR increased (Investigations) | 4 | 3
Icteric sclera (Eye disorders) | 1 | 0
Impaired liver function (Hepatobiliary disorders) | 0 | 1
Incomplete right bundle branch block (Cardiac disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased platelets (Investigations) | 1 | 0
Increased serum creatinine (Investigations) | 0 | 1
Influenza A virus infection (Infections and infestations) | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0
Interventricular septum rupture (Cardiac disorders) | 1 | 0
Intra-abdominal infection (Infections and infestations) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Ionized calcium decreased (Investigations) | 2 | 1
Ionized calcium increased (Investigations) | 1 | 0
Iron binding capacity decreased (Investigations) | 1 | 1
Iron binding capacity unsaturated decreased (Investigations) | 1 | 0
Iron decreased (Investigations) | 2 | 1
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Jugular catheterisation (Surgical and medical procedures) | 0 | 1
Ketone bodies urine positive (Investigations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lipase increased (Investigations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Localized edema (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Lung infection NOS (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Lymphocyte percentage decreased (Investigations) | 3 | 2
Lymphocytes atypical (Investigations) | 1 | 1
MAP increased (Investigations) | 1 | 0
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 | 2
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 | 3
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Mean cell volume increased (Investigations) | 0 | 1
Mean platelet volume increased (Investigations) | 3 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Metamyelocyte count increased (Investigations) | 0 | 1
Migraine headache (Nervous system disorders) | 0 | 1
Mitral regurgitation (Cardiac disorders) | 1 | 0
Monocyte percentage decreased (Investigations) | 1 | 0
Monocytes increased (Investigations) | 2 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Myelocyte count increased (Investigations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myoclonus (Nervous system disorders) | 1 | 0
NT-proBNP increased (Investigations) | 1 | 0
Nasogastric tube insertion (Surgical and medical procedures) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Nephrostomy tube placement (Surgical and medical procedures) | 0 | 1
Nephrotoxicity (Renal and urinary disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1
Neutrophil percentage increased (Investigations) | 1 | 0
Neutrophils increased (Investigations) | 1 | 1
Nitrite urine present (Investigations) | 2 | 0
Normocytic anemia (Blood and lymphatic system disorders) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Numbness oral (Gastrointestinal disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 2
Oedema of mouth (Gastrointestinal disorders) | 1 | 0
Open spina bifida (Congenital, familial and genetic disorders) | 0 | 1
Opiates positive (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Oxygen saturation low (Investigations) | 1 | 0
PCO2 increased (Investigations) | 1 | 0
PO2 increased (Investigations) | 1 | 0
PTH increased (Investigations) | 1 | 0
Pain oral (Gastrointestinal disorders) | 1 | 0
Pancreas cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Perioral paraesthesia (Gastrointestinal disorders) | 1 | 0
Peripheral neuropathy NOS (Nervous system disorders) | 1 | 1
Platelet count decreased (Investigations) | 2 | 3
Platelet count increased (Investigations) | 0 | 2
Platelets decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion recurrent (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Prealbumin decreased (Investigations) | 3 | 0
Pressure sore (Skin and subcutaneous tissue disorders) | 1 | 0
Progressive renal failure (Renal and urinary disorders) | 1 | 3
Protein total decreased (Investigations) | 1 | 0
Protein total increased (Investigations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 5 | 5
Prothrombin time increased (Investigations) | 3 | 4
Prothrombin time prolonged (Investigations) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pulse decreased (Investigations) | 1 | 0
Red blood cell distribution width increased (Investigations) | 1 | 1
Red blood cell morphology abnormal (Investigations) | 0 | 2
Renal injury (Renal and urinary disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Respiratory infection (Infections and infestations) | 1 | 0
Respiratory rate decreased (Investigations) | 1 | 0
Respiratory rate increased (Investigations) | 1 | 1
Restlessness aggravated (Psychiatric disorders) | 1 | 0
Reticulocyte count increased (Investigations) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Scrotal ulcer (Reproductive system and breast disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 2
Sepsis (Infections and infestations) | 24 | 22
Septic shock (Infections and infestations) | 8 | 2
Septicemia due to Escherichia coli (E. coli) (Infections and infestations) | 1 | 0
Serum calcium decreased (Investigations) | 0 | 1
Serum chloride increased (Investigations) | 2 | 0
Serum creatinine decreased (Investigations) | 0 | 1
Serum creatinine increased (Investigations) | 0 | 1
Serum osmolality increased (Investigations) | 0 | 1
Serum total protein decreased (Investigations) | 3 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus rhythm (Investigations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Specific gravity urine decreased (Investigations) | 0 | 1
Specific gravity urine increased (Investigations) | 1 | 0
Staphylococcus aureus test positive (Investigations) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 2
Sudden death (General disorders) | 0 | 1
TPN (Surgical and medical procedures) | 1 | 0
TSH increased (Investigations) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 3
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Tako-Tsubo cardiomyopathy (Cardiac disorders) | 1 | 0
Thoracentesis (Investigations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrush oral (Infections and infestations) | 1 | 0
Total iron binding capacity decreased (Investigations) | 1 | 0
Tracheo-bronchial secretion excess (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transferrin decreased (Investigations) | 3 | 0
Triglyceride increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 2
Troponin NOS (Investigations) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Unspecified osteomyelitis involving lower leg (Infections and infestations) | 0 | 1
Urinary casts present (Investigations) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urine RBC increased (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Urine bilirubin increased (Investigations) | 1 | 1
Urine calcium oxalate crystal present (Investigations) | 1 | 0
Urine epithelial cells increased (Investigations) | 3 | 0
Urine ketone body present (Investigations) | 1 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 4
Urine red blood cells increased (Investigations) | 1 | 2
Urine white blood cell increased (Investigations) | 1 | 0
Urobilinogen urine increased (Investigations) | 0 | 2
Vena cava filter insertion (Surgical and medical procedures) | 0 | 1
Ventilator associated pneumonia (Infections and infestations) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vitamin B12 increased (Investigations) | 1 | 0
Vitamin D decreased (Investigations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
WBC increased (Investigations) | 1 | 2
Weight increased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 1 | 0
White blood cells urine increased (Investigations) | 2 | 1
White blood cells urine positive (Investigations) | 1 | 0
Zinc decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT01597973/Prot_SAP_000.pdf